CLINICAL TRIAL: NCT03530709
Title: Traditional vs Virtually-integrated Co-management of Children With Medical Complexity Between Complex Care and Community-based Primary Care Providers
Brief Title: Virtually-integrated Co-management Between Complex Care and Community-based Primary Care Providers
Acronym: CoTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-1889
Record Dates: First submitted 2018-04-18; First posted 2018-05-21 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Chronic Illness
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): videoconferencing
  Interventions: Other: videoconferencing
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: videoconferencing — Parents/caregivers will use smartphones to videoconference in their SCC provider during PCP visits
  Arms: Experimental

SUMMARY:
This is a pilot trial to test whether tertiary center-affiliated pediatricians with expertise in medical complexity joining medical visits with patients' community primary care providers is feasible and acceptable. We will also collect data on a range of patient-centered and utilization outcomes to determine effect compared to usual care.

ELIGIBILITY:
Inclusion Criteria: Caregiver of patient seen for co-managed care in Special Care Clinic; caregiver has a smartphone that will accept the technology; PCPs office has wireless internet connection -

Exclusion Criteria: Child is in foster care

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of co-managed visits scheduled that are completed through videoconferencing | 12 months
  To determine the feasibility of scheduled visits that are completed through videoconferencing

SECONDARY OUTCOMES:
Caregiver Perception of integrated care | Baseline, 3 months and 6 months
  Instrument that measures the perception of how well care is integrated. This is a validated, caregiver-reported outcome

OTHER OUTCOMES:
Caregiver Satisfaction with Telehealth | After every telehealth visit (up to 3 visits)
  Adapted validated, caregiver-reported measure of satisfaction with the telehealth visit

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Van Cleave, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No